CLINICAL TRIAL: NCT05888714
Title: Pilot Study for Peripheral Neuromuscular Electrical Stimulation of the Quadriceps Muscle: Healthy or Deprived of Central Nervous System Control
Brief Title: Pilot Study for Peripheral Neuromuscular Electrical Stimulation of the Quadriceps Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Agência Brasileira de Desenvolvimento Industrial (Brazilian Agency For Industrial Development) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 64324122.0.0000.0068
Record Dates: First submitted 2023-04-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injuries; Brain Injuries; Muscle Atrophy
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental FES cycling (Experimental): New medical device combining cycle ergometer use and neuromuscular electrical stimulation (FES cycling)
  Interventions: Device: Experimental FES cycling
- Comparator FES cycling (Active Comparator): Existing medical device combining cycle ergometer use and neuromuscular electrical stimulation (FES cycling)
  Interventions: Device: Comparator FES cycling
- Conventional physical therapy (Active Comparator): Conventional physical therapy.
  Interventions: Other: Conventional physical therapy
- Operators (No Intervention): Operators will evaluate systems usability during interventions.

INTERVENTIONS:
Device: Experimental FES cycling — Using the experimental, new FES cycling device, provide neuromuscular electrical stimulation of the gluteal, quadriceps and hamstring muscles at sufficient intensity to cause muscle contraction and push the cycle ergometer pedals for 30 minutes, for 16 treatment sessions (twice a week, for 8 weeks), in addition to conventional physical therapy for muscle strengthening.
  Arms: Experimental FES cycling
Device: Comparator FES cycling — Using the comparator, marketed FES cycling device, provide neuromuscular electrical stimulation of the gluteal, quadriceps and hamstring muscles at sufficient intensity to cause muscle contraction and push the cycle ergometer pedals for 30 minutes, for 16 treatment sessions (twice a week, for 8 weeks), in addition to conventional physical therapy for muscle strengthening.
  Arms: Comparator FES cycling
Other: Conventional physical therapy — Conventional physical therapy for muscle strengthening, for 16 treatment sessions (twice a week, for 8 weeks).
  Arms: Conventional physical therapy

SUMMARY:
Feasibility study of a new medical device that will evaluate the usability and effectiveness of a cycle ergometer device associated with neuromuscular electrical stimulation (FES cycling). The study's objective is to evaluate the effect of the application of functional electrical stimulation of the new device on participants' quadriceps muscle strength in comparison to a medical device with similar characteristics and to a control group. Secondarily, the study will compare the usability of the two medical devices as evaluated by the participants and the therapists who apply the treatment, as well as the participants' satisfaction with the treatment, identifying possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury, brain injury or acquired muscle weakness
* Managed chronic diseases
* No contraindications to the practice of physical exercise
* Ability to communicate in oral and written Portuguese

Exclusion Criteria:

* Amputation of lower limbs at any level
* Unstable or acute fractures of lower limbs
* Contraindication for the practice of physical activity
* Open wounds in the lower limbs
* Consent withdraw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in knee joint extensors peak torque (Newton-Meters) | Change from baseline knee joint extensors peak torque at end of intervention, completed 8 weeks after initiation
  Quadriceps muscle strength, measured by isokinetic dynamometry
Change in knee joint flexors peak torque (Newton-Meters) | Change from baseline knee joint flexors peak torque at end of intervention, completed 8 weeks after initiation
  Quadriceps muscle strength, measured by isokinetic dynamometry
Change in thigh perimeter (centimeters) | Change from baseline thigh perimeter at end of intervention, completed 8 weeks after initiation
  Quadriceps muscle integrity, measured by thigh volumetry
Change in rectus femoris thickness (centimeters) | Change from baseline rectus femoris thickness at end of intervention, completed 8 weeks after initiation
  Rectus femoris muscle structural integrity, measured by ultrasound
Change in vastus intermedius thickness (centimeters) | Change from baseline vastus intermedius thickness at end of intervention, completed 8 weeks after initiation
  Vastus intermedius muscle structural integrity, measured by ultrasound

SECONDARY OUTCOMES:
System Usability Score | System usability at end of intervention, completed 8 weeks after initiation
  Systems usability, measured by self-referred survey (0-100, the higher the score, the better the outcome)
Patients Perception of Treatment Outcomes Score | Patients perception of treatment outcomes at end of intervention, completed 8 weeks after initiation
  Satisfaction, measured by self-referred survey (6-30, the higher the score, the better the outcome)
Adverse effects inventory | Adverse effects at end of each treatment session with the assigned intervention, completed 30min after session initiation
  Qualitative evaluation of adverse effects, if any

CONTACTS AND LOCATIONS:
Overall Officials: Linamara R. Battistella, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Medicina Física e Reabilitação, Hospital das Clínicas, Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Result] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Result] Scheuringer M, Grill E, Boldt C, Mittrach R, Mullner P, Stucki G. Systematic review of measures and their concepts used in published studies focusing on rehabilitation in the acute hospital and in early post-acute rehabilitation facilities. Disabil Rehabil. 2005 Apr 8-22;27(7-8):419-29. doi: 10.1080/09638280400014089. PMID 16040545
- [Result] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Result] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Result] Stoll T, Brach M, Huber EO, Scheuringer M, Schwarzkopf SR, Konstanjsek N, Stucki G. ICF Core Set for patients with musculoskeletal conditions in the acute hospital. Disabil Rehabil. 2005 Apr 8-22;27(7-8):381-7. doi: 10.1080/09638280400013990. PMID 16040540
- [Result] van der Schaaf M, Beelen A, Dongelmans DA, Vroom MB, Nollet F. Poor functional recovery after a critical illness: a longitudinal study. J Rehabil Med. 2009 Nov;41(13):1041-8. doi: 10.2340/16501977-0443. PMID 19893999
- [Result] Martin UJ, Hincapie L, Nimchuk M, Gaughan J, Criner GJ. Impact of whole-body rehabilitation in patients receiving chronic mechanical ventilation. Crit Care Med. 2005 Oct;33(10):2259-65. doi: 10.1097/01.ccm.0000181730.02238.9b. PMID 16215380
- [Result] Garnacho-Montero J, Amaya-Villar R, Garcia-Garmendia JL, Madrazo-Osuna J, Ortiz-Leyba C. Effect of critical illness polyneuropathy on the withdrawal from mechanical ventilation and the length of stay in septic patients. Crit Care Med. 2005 Feb;33(2):349-54. doi: 10.1097/01.ccm.0000153521.41848.7e. PMID 15699838
- [Result] Dittmer DK, Teasell R. Complications of immobilization and bed rest. Part 1: Musculoskeletal and cardiovascular complications. Can Fam Physician. 1993 Jun;39:1428-32, 1435-7. PMID 8324411
- [Result] Pinheiro AR, Christofoletti G. Motor physical therapy in hospitalized patients in an intensive care unit: a systematic review. Rev Bras Ter Intensiva. 2012 Jun;24(2):188-96. English, Portuguese. PMID 23917769
- [Result] Maddocks M, Armstrong S, Wilcock A. Exercise as a supportive therapy in incurable cancer: exploring patient preferences. Psychooncology. 2011 Feb;20(2):173-8. doi: 10.1002/pon.1720. PMID 20333769